CLINICAL TRIAL: NCT03771651
Title: A Surgical Window Pilot Investigation of Short Term Aspirin on the Biologic and Immunologic Changes of the Fallopian Tube
Brief Title: Short Term Aspirin on the Biologic and Immunologic Changes of the Fallopian Tube
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9955
Record Dates: First submitted 2018-12-07; First posted 2018-12-11 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Fallopian Tube Cancer; Fallopian Tube Infection
MeSH Terms: conditions — Fallopian Tube Neoplasms | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Aspirin (Experimental): Subjects will take 81mg tablets of aspirin daily for 14 days prior to surgery for removal of fallopian tubes.
  Interventions: Drug: Aspirin 81 mg

INTERVENTIONS:
Drug: Aspirin 81 mg — Subjects will take aspirin daily for 14 days leading up to surgery to determine whether it impacts inflammation of fallopian tubes.

SUMMARY:
This study will evaluate the impact of low dose aspirin on normal fallopian tube fimbriae in women who have surgery to have their fallopian tubes removed. Participants will take a low dose of aspirin for 2 weeks before their surgery. A portion of the removed fallopian tubes will also be collected for future research and routine pathology purposes.

DETAILED DESCRIPTION:
Subjects in this study will receive low dose aspirin for 14 days before undergoing surgery to remove fallopian tubes removed to determine whether aspirin decreases inflammation in the fallopian tube. Subjects will also submit blood samples at their initial visit with their oncologist, at the time of surgery and at the pre-operative visit to measure inflammation markers and blood counts. A portion of the subject's fallopian tube will be collected for future research studies.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing gynecologic surgery for presumed benign indications that includes the removal of their fallopian tubes. This may include sterilization procedures, hysterectomy or partial or full adnexectomy.
* Eligible women will have fulfilled their childbearing desires
* Age > 21 Considered low risk for prevalent fallopian tube cancer (not undergoing risk reducing surgery for a known BRCA mutation or other known hereditary predisposition syndrome, family history of ovarian cancer in a first degree relative.

Exclusion Criteria:

* Males
* Women who have presumed or known gynecologic cancer
* Women less than 21 years of age
* Women currently on either regular aspirin therapy, non-steroidal anti-inflammatory drugs (NSAIDS), acetaminophen or chronic steroidal anti-inflammatory medications.
* Women with known bleeding diathesis or bleeding disorder.
* Women who do not consent for removal of both fallopian tubes.
* Women with a history of gastritis or peptic ulcer disease requiring treatment. (Patients with a history of occasional H1 or H2 blocker use for gastro esophageal reflux disease are NOT excluded).
* Women with reported aspirin or NSAID allergy
* Women with asthma and/or nasal polyps

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Number of subjects who exhibited alterations in the fallopian tube immune microenvironment | 5 years
  Immuno-cellular assays and percentages of specific immune cells will be compared to control tissue samples.
Number of subjects who exhibited less carcinogenic potential than control specimens | 5 years
  Ciliate cells from specimens will be isolated and the number of colony forming units will be compared to control samples.
Number of subjects who exhibited changes in transcriptome profile compared to control specimens | 5 years
  Normal fallopian tube fibria will be compared to ovarian cancer specimens to identify novel biomarkers for diagnosis, targets for prevention and better treatment strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Holman, Principal Investigator — Stephenson Cancer Center, University of Oklahoma Health Sciences Center
Locations (1):
- Stephenson Cancer Center, University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No